CLINICAL TRIAL: NCT00642967
Title: A Single Arm, Open Label, French Multi-centre Study to Assess the Maintenance of Hemoglobin Levels With Once Monthly Subcutaneous Administration of C.E.R.A. (Continuous Erythropoietin Receptor Activator) in Patients With Chronic Kidney Disease Not on Dialysis
Brief Title: A Study of Subcutaneous Mircera for the Maintenance Treatment of Anemia in Participants With Chronic Kidney Disease Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21146; 2007-005757-28 (EudraCT Number)
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Methoxy Polyethylene Glycol-epoetin Beta (Experimental): Participants will receive subcutaneous methoxy polyethylene glycol-epoetin beta every 4 weeks for a total of 48 weeks in this single-arm study. The first dose of 120 or 200 micrograms (mcg) will be determined based on the previous dose of epoetin or darbepoetin received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within the target range.
  Interventions: Drug: Methoxy Polyethylene Glycol-epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-epoetin Beta — Methoxy polyethylene glycol-epoetin beta will be administered subcutaneously every 4 weeks for a total of 48 weeks in this single-arm study. The first dose of 120 or 200 mcg will be determined based on the previous dose of epoetin or darbepoetin received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within the target range.
  Other Names: Mircera; C.E.R.A

SUMMARY:
This single arm study will assess the efficacy and safety of monthly administration of subcutaneous methoxy polyethylene glycol-epoetin beta (Mircera) when administered for the maintenance of hemoglobin levels in participants with chronic renal anemia, not on dialysis. Participants currently receiving treatment with subcutaneous epoetin or darbepoetin alfa will receive monthly subcutaneous injections of methoxy polyethylene glycol-epoetin beta, with the starting dose (120 or 200 micrograms) calculated from the last weekly dose of epoetin beta or darbepoetin alfa previously administered.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease stage 3 or 4, with chronic renal anemia, not requiring dialysis;
* continuous stable subcutaneous maintenance Erythropoietin-Stimulating Agent (ESA) therapy during previous month.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* significant acute or chronic bleeding;
* poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients maintaining average Hb concentration within target range of 10-12g/dL during evaluation period | Weeks 16-24

SECONDARY OUTCOMES:
Mean change in Hb concentration | Between reference and Efficacy Evaluation Period
Mean time spent in Hb range | Weeks 16-24
% patients maintaining Hb concentration within target range; % patients requiring dose adjustments; incidence of RBC transfusions | Weeks 16-48
AEs, lab parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- France (63):
  - Aix-en-Provence
  - Angers
  - Annonay
  - Avignon
  - Bastia
  - Beauvais
  - Besançon
  - Bois-Guillaume
  - Bordeaux
  - Boulogne-sur-Mer
  - Bourg-en-Bresse
  - Bourges
  - Brest
  - Caen
  - Chalon-sur-Saône
  - Chartres
  - Cherbourg Octeville
  - Cholet
  - Clermont-Ferrand
  - Colmar
  - Creil
  - Créteil
  - Dieppe
  - Évreux
  - Greize
  - Harfleur
  - La Garenne-Colombes
  - La Tronche
  - Le Havre
  - Le Mans
  - Lille
  - Limoges
  - Lyon
  - Maubeuge
  - Metz
  - Metz-Tessy
  - Montluçon
  - Montpellier
  - Nancy
  - Nice
  - Nîmes
  - Orléans
  - Paris
  - Pierre-Bénite
  - Poitiers
  - Quimper
  - Roubaix
  - Saint-Brieuc
  - Saint-Laurent-du-Var
  - Saint-Lô
  - Saint-Michel
  - Saint-Nazaire
  - Salouël
  - Sens
  - St-Malo
  - Strasbourg
  - Suresnes
  - Thionville
  - Toulouse
  - Tournan-en-Brie
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes